CLINICAL TRIAL: NCT02892422
Title: Interventional, Open-label, Flexible-dose, Long-term Safety Study of Lu AF35700 in Adult Patients With Schizophrenia
Brief Title: Flexible-dose, Long-term Safety Study of Lu AF35700 in Adult Patients With Schizophrenia
Acronym: Debut
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16159B; 2015-003284-11 (EudraCT Number)
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lu AF35700

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flexible-dose of Lu AF35700 (Experimental)
  Interventions: Drug: Lu AF35700

INTERVENTIONS:
Drug: Lu AF35700 — Flexible-dose of Lu AF35700, 10 or 20 mg/day, tablets, orally.
  From Day 8, the daily dose can be increased to 20mg. Thereafter, the daily dose can be adjusted (decreased to 10mg or following a decrease, increased to 20mg/day)
  Patients who completed the 16159A study, only, can be switched to a weekly 70 mg Lu AF35700 dosing regimen (tablets, orally, once weekly) after 8 weeks in this study

SUMMARY:
To evaluate the safety and tolerability of the long-term treatment with Lu AF35700.

DETAILED DESCRIPTION:
Safety study in patients with schizophrenia who have participated and completed a study investigating Lu AF35700 including Studies 16159A and 16323A. Or in patients with schizophrenia for whom a switch of antipsychotic treatment can be potentially beneficial according to the investigator's clinical judgement.

ELIGIBILITY:
Inclusion Criteria:

- For 16159A-patients

* The patient has completed Study 16159A.
* The patient is able to read and understand the Informed Consent Form.
* The patient has signed the Informed Consent Form specific for Study 16159B.
* The patient can potentially benefit from 52-week treatment with Lu AF35700 according to the investigator's clinical judgement.

For 16323A-patients

* The patient has completed the dosing period of Study 16323A.
* The patient is able to read and understand the Informed Consent Form.
* The patient has signed the Informed Consent Form specific Study 16159B.
* The patient has a confirmed diagnosis of schizophrenia according to DSM-5™.
* The patient can potentially benefit from 52-week treatment with Lu AF35700 according to the investigator's clinical judgement.

For Other Patients

* The patient has schizophrenia, diagnosed according to DSM-5™.
* The patient is a man or woman, aged ≥18 years.
* The patient has been prescribed oral antipsychotic treatment at the recommended dose range as stated in the summary of product characteristics or equivalent label for 6 weeks prior to the Screening Visit.
* The patient has a PANSS total score ≥60 and ≤90 at Screening and Baseline Visits.
* The patient has a Clinical Global Impression - Severity of Illness (CGI-S) score ≤4.
* The patient is in need of a change in the current antipsychotic treatment and, according to the investigator's clinical judgement, the patient can potentially benefit from a switch to another treatment including, but not limited to, any of the following reasons:

  * lack of adequate response to his or her current antipsychotic medication;
  * poor tolerability to his or her current antipsychotic medication;
  * unwillingness of the patient to adhere to his or her current antipsychotic medication.

Exclusion Criteria:

- For 16159A-patients

* The patient has been diagnosed with a primary psychiatric disorder other than schizophrenia during Study 16159A.
* The patient, in the opinion of the investigator, is at significant risk of suicide, or: Answers "Yes" to any question on the Suicidal Behaviour section of the Columbia-Suicide Severity Rating Scale (C-SSRS), OR Answers "Yes" to questions 4 and 5 on the Suicidal Ideation section of the C-SSRS

For 16323A-patients

* The patient has been diagnosed with a primary psychiatric disorder other than schizophrenia during Study 16323A.
* The patient, in the opinion of the investigator, is at significant risk of suicide, or: Answers "Yes" to any question on the Suicidal Behaviour section of the C-SSRS, OR Answers "Yes" to questions 4 and 5 on the Suicidal Ideation section of the C-SSRS

For Other Patients

* The patient has any current psychiatric disorder (DSM-5™ criteria) other than schizophrenia established as the primary diagnosis.
* The patient is experiencing acute exacerbation of psychotic symptoms at the Screening Visit, between the Screening and Baseline Visits or at the Baseline Visit.
* The patient is treated with clozapine at the time of the Screening Visit.
* The patient has a substance use disorder (except nicotine) which according to the investigator's judgment may compromise the patient's ability to comply with the study procedures, or preclude the benefits of the study medication.
* The patient, in the opinion of the investigator, is at significant risk of suicide, or: Answers "Yes" to any question on the Suicidal Behaviour section of the C-SSRS, OR Answers "Yes" to questions 4 and 5 on the Suicidal Ideation section of the C-SSRS

Other protocol defined inclusion and exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (102):
- United States (32):
  - US1018, Bellflower, California
  - US1062, Costa Mesa, California
  - US1463, Culver City, California
  - US1399, Escondido, California
  - US1104, Garden Grove, California
  - US1114, National City, California
  - US1459, Oceanside, California
  - US1368, Orange, California
  - US1391, San Bernardino, California
  - US1392, Torrance, California
  - US1318, Lauderhill, Florida
  - US1130, Miami, Florida
  - US1129, North Miami, Florida
  - US1402, Oakland Park, Florida
  - US1403, Atlanta, Georgia
  - US1009, Atlanta, Georgia
  - US1046, Chicago, Illinois
  - US1423, Hoffman Estates, Illinois
  - US1398, Shreveport, Louisiana
  - US1404, Shreveport, Louisiana
  - US1086, Flowood, Mississippi
  - US1444, Las Vegas, Nevada
  - US1426, Berlin, New Jersey
  - US1244, Fresh Meadows, New York
  - US1394, New York, New York
  - US1416, New York, New York
  - US1171, Rochester, New York
  - US1190, Staten Island, New York
  - US1390, Charlotte, North Carolina
  - US1124, Norristown, Pennsylvania
  - US1451, Austin, Texas
  - US1065, Dallas, Texas
- Bulgaria (9):
  - BG1030, Burgas
  - BG1028, Kazanlak
  - BG1003, Lovech
  - BG1008, Plovdiv
  - BG1024, Sofia
  - BG1026, Sofia
  - BG1034, Varna
  - BG1029, Veliko Tarnovo
  - BG1027, Vratsa
- CA1029, Penticton, Canada
- Czechia (4):
  - CZ1023, Brno
  - CZ1032, Brno
  - CZ1013, Lnáře
  - CZ1038, Prague
- EE1007, Tallinn, Estonia
- Mexico (8):
  - MX1024, Durango
  - MX1011, Guadalajara
  - MX1021, Guadalajara
  - MX1022, Guadalajara
  - MX1020, Mexico City
  - MX1005, Monterrey
  - MX1007, Monterrey
  - MX1015, Monterrey
- Poland (5):
  - PL1043, Bialystok
  - PL1060, Lodz
  - PL1058, Pruszcz Gdański
  - PL1059, Torun
  - PL1051, Wroclaw
- RO1024, Bucharest, Romania
- Russia (14):
  - RU1009, Arkhangelsk
  - RU1021, Gatchina
  - RU1006, Moscow
  - RU1051, Moscow
  - RU1055, Moscow
  - RU1053, Roshchino
  - RU1023, Saint Petersburg
  - RU1028, Saint Petersburg
  - RU1030, Saint Petersburg
  - RU1031, Saint Petersburg
  - RU1049, Saint Petersburg
  - RU1052, Saint Petersburg
  - RU1056, Saint Petersburg
  - RU1050, Yaroslavl
- Serbia (8):
  - RS1008, Belgrade
  - RS1010, Belgrade
  - RS1012, Belgrade
  - RS1001, Kovin
  - RS1011, Kragujevac
  - RS1016, Kragujevac
  - RS1017, Kragujevac
  - RS1009, Novi Kneževac
- Slovakia (3):
  - SK1014, Bratislava
  - SK1024, Bratislava
  - SK1026, Zlaté Moravce
- Spain (3):
  - ES1047, Barcelona
  - ES1008, Málaga
  - ES1048, Oviedo
- Ukraine (13):
  - UA1017, Kharkiv
  - UA1035, Kharkiv
  - UA1029, Kherson
  - UA1027, Kiev
  - UA1028, Kiev
  - UA1030, Kiev
  - UA1031, Kiev
  - UA1033, Lviv
  - UA1019, Odesa
  - UA1020, Odesa
  - UA1032, Oleksandrivka
  - UA1001, Poltava
  - UA1036, Vinnitsa

REFERENCES:
- [Derived] Kane JM, Kinon BJ, Forray C, Such P, Mittoux A, Lemming OM, Hertel P, Howes OD; DayBreak and Debut study investigators. Efficacy and safety of Lu AF35700 in treatment-resistant schizophrenia: A randomized, active-controlled trial with open-label extension. Schizophr Res. 2022 Oct;248:271-278. doi: 10.1016/j.schres.2022.09.012. Epub 2022 Sep 14. PMID 36115192

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had completed either study 16159A or 16323A were enrolled. Participants from study 16323A were excluded from the "all patients treated dataset" and from the "full analysis dataset".
Groups:
- Lu AF35700 Flexible-dose: Lu AF35700: Flexible-dose of Lu AF35700, 10 or 20 mg/day, tablets, orally. From Day 8, the daily dose can be increased to 20mg. Thereafter, the daily dose can be adjusted (decreased to 10mg or following a decrease, increased to 20mg/day) Patients who completed the 16159A study, only, can be switched to a weekly 70 mg Lu AF35700 dosing regimen (tablets, orally, once weekly) after 8 weeks in this study
Period: Overall Study
Arm/Group | Lu AF35700 Flexible-dose
Started | 528 (528 participants were enrolled, 524 from study 16159A and 4 from study 16323A)
Completed | 318
Not Completed | 210
Not completed — Enrolled not treated | 4
Not completed — Adverse Event | 38
Not completed — Lack of Efficacy | 32
Not completed — Non-compliance with study drug | 11
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 56
Not completed — Lost to Follow-up | 5
Not completed — sponsor information 16159A results | 21
Not completed — withdrawal of consent | 13
Not completed — exclusion criteria met | 3
Not completed — moving elsewhere | 4
Not completed — non-compliance | 10
Not completed — patient legally incapable | 1
Not completed — patient decision | 7
Not completed — Investigator decision | 1

BASELINE CHARACTERISTICS:
Population: Participants who had completed either study 16159A or 16323A were enrolled. Participants from study 16323A were excluded from the "all patients treated dataset" and from the "full analysis dataset".
Arm/Group | Flexible-dose of Lu AF35700
Number analyzed (Participants) | 528
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220
  Male | 308
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 63
  White | 412
  More than one race | 0
  Unknown or Not Reported | 51
Region of Enrollment [Number; unit: participants]
  Romania | 3
  United States | 98
  Czechia | 11
  Ukraine | 48
  Russia | 112
  Spain | 3
  Canada | 3
  Poland | 19
  Mexico | 57
  Slovakia | 8
  Bulgaria | 107
  Serbia | 43
  Estonia | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: Based on the safety assessments (e.g. clinical safety laboratory tests, vital signs, weight, waist circumference and ECG)
Time Frame: From dosing to end of study (57 weeks)
Population: Participants from study 16323A were excluded from the "all patients treated dataset" and from the "full analysis dataset".
Measure: Count of Participants; unit: Participants
Arm/Group | Flexible-dose of Lu AF35700
Number analyzed (Participants) | 524
Participants | 289

ADVERSE EVENTS:
Time Frame: 57 weeks
Groups:
- Lu AF35700 Flexible-dose: Lu AF35700: Flexible-dose of Lu AF35700, 10 or 20 mg/day, tablets, orally.
Arm/Group | Lu AF35700 Flexible-dose
All-Cause Mortality (participants affected / at risk) | 0/524
Serious Adverse Events (participants affected / at risk) | 28/524
Other Adverse Events (participants affected / at risk) | 43/524
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lu AF35700 Flexible-dose (N=524)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 2 (2)
Coma (Nervous system disorders) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Disinhibition (Psychiatric disorders) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 3 (3)
Schizophrenia (Psychiatric disorders) | 16 (19)
Suicide attempt (Psychiatric disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lu AF35700 Flexible-dose (N=524)
Headache (Nervous system disorders) | 43 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-05-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT02892422/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT02892422/SAP_001.pdf